CLINICAL TRIAL: NCT00565513
Title: Cryptorchidism: Impact of in Utero Exposure to Xenobiotics With Hormonal Action and Multidisciplinary
Brief Title: Cryptorchidism: Impact of in Utero Exposure to Xenobiotics With Hormonal Action
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Cynthia GIRAN, Département de la Recherche Clinique et de l'Innovation
Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PHRC 2001
Record Dates: First submitted 2007-11-29; First posted 2007-11-30 (Estimated); Last update posted 2007-11-30 (Estimated); Status verified 2007-11

CONDITIONS: Cryptorchidism
MeSH Terms: conditions — Cryptorchidism | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Other): cord blood and maternal milk tests
  Interventions: Procedure: blood test

INTERVENTIONS:
Procedure: blood test — cord blood and maternal milk test

SUMMARY:
We studied prospectively the incidence of cryptorchidism in Nice area. We tightly matched each affected child (n=95) with 2 healthy controls (n=188) and assessed risk factors for cryptorchidism focussing on prenatal exposure (cord blood and maternal milk) to endocrine disruptors known to affect testis migration, searching for correlations with cryptorchid status

DETAILED DESCRIPTION:
Since fetal exposure to anti-androgenic and/or estrogenic compounds is deleterious to animal reproduction, such exposure could be harmful to human fetus as well. Data are scarce on human exposure and the occurrence of cryptorchidism.

DESIGN: From 2002 to 2005, we performed a prospective case-control study to assess the incidence of cryptorchidism and fetal exposure to selected chemicals in newborn boys in Nice area. This study was approved by the ethical board of our institution. Out of 6246 live births at or after 34 weeks of gestational age and born at 2 maternity wards (University hospital of Nice and General Hospital of Grasse), 102 boys were diagnosed with cryptorchidism. After informed parental consent, 95 were included in this study, along with 188 tightly matched controls. Cord blood was collected at birth, as well as maternal milk from nursing mothers. Lifestyle and job questionnaires were filled by parents. Children were re-examined at 3 and 12 months of age to assess possible secondary testis migration, or confirm their control status.

151 cord bloods (67 cryptorchid, 84 controls) and 125 maternal milks (56 for cryptorchid boys and 69 for controls) were collected and screened for xenobiotics, including DDE, PCBs, and dibutylphthalate (and metabolite monobutylphthalate -mBP). We established scores of exposure in colostrum and studied possible relationships between exposure and cryptorchidism. We also measured hormonal status on cord blood including AMH and inhibin concentrations.

RESULTS: The incidence of cryptorchidism was 1.6% at birth, similar in Nice and Grasse, and 0.8% at 3 months of age. Xenobiotic measurements in cord blood and milk showed universal exposure in our population. Median concentrations in maternal milk were higher though not significantly in cryptorchid vs controls: DDE 119.4 vs 80 ng/g of fat, ΣPCB 206.3 vs 166.8 ng/g of fat, mBP 17.3 vs 10.3 ng/g of milk. Cryptorchid boys were more likely to be classified in the most contaminated groups for ΣPCBs (57.1% vs 39.1% p=0.045), DDE (53.6 vs 36.2% p=0.037) and to a lesser degree mBP (58.1 vs 40%, p=0.13). This was also true for the composite score using DDE and ΣPCBs (30.4 vs 21.7%, p=0.05). Last, the odds ratio for cryptorchidism at birth was increased for the highest score of: DDE: 2.03 (p=0.05, 95%CI 0.99-4.17); ΣPCB 2.07 (p=0.046, 95%CI 1.01-4.25); composite score without phthalates 2.41 (p=0.06, 95%CI 0.96-6.1) vs the lowest score of those components.

CONCLUSIONS: The incidence of cryptorchidism at birth of 1.6% is similar to other populations. Our results support an association between fetal exposure to DDE, PCBs and possibly mBP, and the occurrence of cryptorchidism at birth. Higher concentrations in milk could be a marker of higher exposure or for an impaired detoxification pattern in genetically predisposed individuals. Long term follow up of our cohort is planned to screen cryptorchid and control boys for low sperm count, infertility and testis cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women having given birth to a boy at University hospital of Nice or Général hospital of Grasse

Exclusion Criteria:

* parents who don't signed consent

Max Age: 1 Year | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 283 (Actual)
Dates: Start 2002-04; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Neonatal examination for the diagnosis of undescended testis (cryptorchidism) | At birth, 3 and 12 month of age

SECONDARY OUTCOMES:
Measurement of xenobiotic concentrations in cord blood and maternal milk in cryptorchid and control boys Parental questionnaires: demographic information, lifestyle, job exposure Pregnancy, delivery and neonatal other information | At birth

CONTACTS AND LOCATIONS:
Overall Officials: Françoise BRUCKER-DAVIS, Doctor, Principal Investigator — Department of Endocrinology of University Hospital of Nice